CLINICAL TRIAL: NCT03541590
Title: Ultrasound-guided Percutaneous Biliary Drainage With Primary Metal Implantation by Endoscopic Luminal Guidance in Patients With Malignant Extrahepatic Bile Duct Obstruction
Brief Title: Ultrasound-guided Percutaneous Biliary Drainage With Primary Metal Implantation by Endoscopic Luminal Guidance
Status: Completed | Type: Observational
Sponsor: Theresienkrankenhaus und St. Hedwig-Klinik GmbH (Other)
Responsible Party: Principal Investigator, Daniel Schmitz, Principal investigator, Theresienkrankenhaus und St. Hedwig-Klinik GmbH
Other Study IDs: PTBD retro 001
Record Dates: First submitted 2018-04-23; First posted 2018-05-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Bile Duct Obstruction, Extrahepatic
Keywords: percutaneous biliary drainage
MeSH Terms: conditions — Cholestasis, Extrahepatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Percutaneous transhepatic biliary drainage — When ERCPs failed or was not possible to be performed due to an altered anatomy in patients with malignant extrahepatic bile duct obstruction, PTBD was performed next in all patients. Percutaneous bile duct puncture was guided by Color Doppler ultrasound. The further procedure was guided by fluoroscopy. A self-expandable metal stent (SEMS) was inserted into the obstructed bile duct by endoscopic luminal guidance in the first session. After successful SEMS implantation, the percutaneous external catheter was removed at the end of the procedure.

SUMMARY:
In a recently published meta-analysis (Sharaiha, Gastrointestinal Endoscopy, 2017), it is reported that percutaneous transhepatic biliary drainage (PTBD) is less clinical successful, causes more adverse events and needs more re-interventions than endoscopic ultrasound guided biliary drainage (EUBD) in patients with malignant, extrahepatic bile duct obstruction. The conclusion was, that EUBD should be prefered in this clinical setting in future.

An improved technique of PTBD may provide better results for coming comparative studies.

The investigators of this retrospective study therefore analyzed all PTBDs that were performed in a period of nine years in a tertiary referral hospital. In this cohort, the analysis focused on PTBDs with primary metal stent implantation by endoscopic luminal guidance.

DETAILED DESCRIPTION:
When Endoscopic Retrograde Cholangiopancreaticography (ERCP) is not successful or is not possible to be performed due to anatomical reasons (altered anatomy after abdominal surgery) in patients with malignant extrahepatic bile duct obstruction, an alternative method is necessary for biliary drainage. In a recently published meta-analysis (Sharaiha, Gastrointestinal Endoscopy, 2017), it is reported that percutaneous transhepatic biliary drainage (PTBD) is less clinical successful, causes more adverse events and needs more re-interventions than endoscopic ultrasound guided biliary drainage (EUBD) in patients with malignant, extrahepatic bile duct obstruction. The conclusion was, that EUBD should be prefered in this clinical setting in future.

An improved technique of PTBD may provide better results for coming comparative studies.

The investigators of this retrospective study therefore analyzed all PTBDs that were performed in a period of nine years in a tertiary referral hospital. In this cohort, the analysis focused on PTBDs with primary metal stent implantation by endoscopic luminal guidance considering technical and clinical success, access route, procedure time, fluoroscopic time, radiation exposure, adverse events and survival probability in an observation time of six months.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* not curatively operable, malignant disease with proximal or distal bile duct obstruction
* elevated serum bilirubin level and/or elevated alkaline phosphatase to at least a twofold degree
* histologically verified diagnosis
* at least one cross-sectional imaging method like computed tomography or magnetic resonance imaging of the abdomen has to be performed

Exclusion Criteria:

* uncorrectable coagulopathy (prothrombin time < 50%, platelet count < 50.000/nl, partial thromboplastin time (PTT) > 50 sec.
* advanced tumor disease with limited life expectancy (< 1 month)
* diffuse liver metastasis
* pregnant or breast feeding women
* potentially curatively, operable, malignant bile duct obstruction
* diseases which can be cured by chemotherapy (for example aggressive non Hodgkin-lymphoma).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients which met the mentioned inclusion and exclusion criteria were enrolled in the study consecutively
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2008-12-01 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
technical success | 1 minute after injection of a radiocontrast agent into the expanded metal stent
  metal stent was implanted successfully bridging the tumor stenosis

SECONDARY OUTCOMES:
clinical success | 7 days
  decrease of Serum Bilirubin level >50%
adverse events | Up to 30 days after the intervention
  the report of any adverse events after the procedure, grading of adverse events according to the ASGE lexicon's severity grading system
re-interventions | 6 months
  Number of re-interventions (ERCP or PTCD) that are necessary after successful PTBD (for example due to stent migration or stent occlusion)
overall survival | 2 years
  death in the follow up afterperformed PTBD

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Rudi, Prof.Dr.med., Study Director — Theresienkrankenhaus und St.Hedwigsklinik GmbH
Locations (1):
- Tertiary referral hospital: Theresienkrankenhaus und St. Hedwig Hospital, Academic, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharaiha RZ, Khan MA, Kamal F, Tyberg A, Tombazzi CR, Ali B, Tombazzi C, Kahaleh M. Efficacy and safety of EUS-guided biliary drainage in comparison with percutaneous biliary drainage when ERCP fails: a systematic review and meta-analysis. Gastrointest Endosc. 2017 May;85(5):904-914. doi: 10.1016/j.gie.2016.12.023. Epub 2017 Jan 4. PMID 28063840
- [Background] Schmitz D, Grosse A, Hallscheidt P, Roseneck A, Niemeyer J, Rudi J. Color Doppler ultrasound-guided PTBD with and without metal stent implantation by endoscopic control: prospective success and early adverse event rates. Z Gastroenterol. 2015 Nov;53(11):1255-60. doi: 10.1055/s-0041-104225. Epub 2015 Nov 12. PMID 26562399
- [Background] Bapaye A, Dubale N, Aher A. Comparison of endosonography-guided vs. percutaneous biliary stenting when papilla is inaccessible for ERCP. United European Gastroenterol J. 2013 Aug;1(4):285-93. doi: 10.1177/2050640613490928. PMID 24917973
- [Background] Artifon EL, Aparicio D, Paione JB, Lo SK, Bordini A, Rabello C, Otoch JP, Gupta K. Biliary drainage in patients with unresectable, malignant obstruction where ERCP fails: endoscopic ultrasonography-guided choledochoduodenostomy versus percutaneous drainage. J Clin Gastroenterol. 2012 Oct;46(9):768-74. doi: 10.1097/MCG.0b013e31825f264c. PMID 22810111
- [Background] Khashab MA, Valeshabad AK, Afghani E, Singh VK, Kumbhari V, Messallam A, Saxena P, El Zein M, Lennon AM, Canto MI, Kalloo AN. A comparative evaluation of EUS-guided biliary drainage and percutaneous drainage in patients with distal malignant biliary obstruction and failed ERCP. Dig Dis Sci. 2015 Feb;60(2):557-65. doi: 10.1007/s10620-014-3300-6. Epub 2014 Aug 1. PMID 25081224
- [Background] Sharaiha RZ, Kumta NA, Desai AP, DeFilippis EM, Gabr M, Sarkisian AM, Salgado S, Millman J, Benvenuto A, Cohen M, Tyberg A, Gaidhane M, Kahaleh M. Endoscopic ultrasound-guided biliary drainage versus percutaneous transhepatic biliary drainage: predictors of successful outcome in patients who fail endoscopic retrograde cholangiopancreatography. Surg Endosc. 2016 Dec;30(12):5500-5505. doi: 10.1007/s00464-016-4913-y. Epub 2016 Apr 29. PMID 27129552
- [Background] Lee TH, Choi JH, Park do H, Song TJ, Kim DU, Paik WH, Hwangbo Y, Lee SS, Seo DW, Lee SK, Kim MH. Similar Efficacies of Endoscopic Ultrasound-guided Transmural and Percutaneous Drainage for Malignant Distal Biliary Obstruction. Clin Gastroenterol Hepatol. 2016 Jul;14(7):1011-1019.e3. doi: 10.1016/j.cgh.2015.12.032. Epub 2015 Dec 31. PMID 26748220
- [Background] Sportes A, Camus M, Greget M, Leblanc S, Coriat R, Hochberger J, Chaussade S, Grabar S, Prat F. Endoscopic ultrasound-guided hepaticogastrostomy versus percutaneous transhepatic drainage for malignant biliary obstruction after failed endoscopic retrograde cholangiopancreatography: a retrospective expertise-based study from two centers. Therap Adv Gastroenterol. 2017 Jun;10(6):483-493. doi: 10.1177/1756283X17702096. Epub 2017 Apr 10. PMID 28567118